CLINICAL TRIAL: NCT04773561
Title: Comparison of Posterior Ocular Changes Between Singleton Pregnancy and Multifetal Pregnancy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Suthasinee Sinawat, Associate Professor, Khon Kaen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HE631549
Record Dates: First submitted 2021-02-25; First posted 2021-02-26 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Twin Pregnancy, Antepartum Condition or Complication; Retinal Vascular; Choroidal Effusion
MeSH Terms: conditions — Choroidal Effusions | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Intervention Model Description: age-stratified sample technique (2 age groups: 24-30 years and 31-37 years)
  ,twin pregnancy:singleton pregnancy:healthy non-pregnant women = 1: 2 : 2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- multifetal pregnancy in the 3rd trimester (Experimental): Corneal tomography, optical coherence tomography and optical coherence tomography angiography were performed in the 3rd trimester, 30-36 weeks of gestational age.
  Interventions: Device: Corneal tomography, optical coherence tomography and optical coherence tomography angiography
- singleton pregnancy in the 3rd trimester (Active Comparator): Corneal tomography, optical coherence tomography and optical coherence tomography angiography were performed in the 3rd trimester, 30-36 weeks of gestational age.
  Interventions: Device: Corneal tomography, optical coherence tomography and optical coherence tomography angiography
- age-stratified healthy non-pregnant women (Active Comparator): Corneal tomography, optical coherence tomography and optical coherence tomography angiography were performed.
  Interventions: Device: Corneal tomography, optical coherence tomography and optical coherence tomography angiography

INTERVENTIONS:
Device: Corneal tomography, optical coherence tomography and optical coherence tomography angiography — Ocular investigations were performed in one time during 30-36 weeks of gestational age. Due to avoidance of diurnal variation, all examinations were done between 10 am - 12 pm.

SUMMARY:
It has been known that a pregnant women undergoes significant anatomical and physiological changes that mainly caused by hormonal and hematologic changes during pregnancy. Due to advance in reproductive medicine, the incidence of multifetal pregnancy was increased to 3% of livebirth. Multifetal pregnancies produce much more physiological changes in the body compared to the singleton pregnancies.

Physiologic ocular changes during pregnancy are the followings

* Melanogenesis of eyelid and facial skin
* Cellular alteration of lacrimal and meibomian gland
* Increased corneal thickness and corneal curvature
* Increased lens thickness
* Increased retinal vascular density
* Increased choroidal thickness Decreased intraocular pressure -

DETAILED DESCRIPTION:
From the literature review, there was only on study of ocular changes in twin pregnancies. Alim et al evaluated the choroidal and retinal thickness in singleton versus twin pregnancies. They included 20 single and 20 twin pregnant women in their 3rd trimester with 20-age-matched healthy non-pregnant women as a control group. They found that there was an increase in choroidal thickness in the 3rd trimester of pregnancies and it was prominent in twin pregnancies. There was a statistically significant difference in choroidal thickness between pregnant and non-pregnant women, but not significant difference between singleton and twin pregnancies. The mean retinal nerve fiber layer thickness was significantly higher in the twin pregnancy group than in the singleton pregnancy group. However, no study of retinal vascular density in twin pregnancies has been published before.

ELIGIBILITY:
Inclusion Criteria:

* 24-37 years
* 30-36 weeks of gestational age
* clear ocular media
* written informed consent

Exclusion Criteria:

* high risk pregnancies such as pre-eclampsia, gestational diabetic mellitus and asthma
* history of refractive error, spherical equivalent > 3 diopters
* history of retinal diseases such as central serous chorioretinopathy and retinal vascular occlusion
* history of intraocular inflammation or endophthalmitis
* history of intraocular laser treatment
* history of intraocular surgery

Ages: 24 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 166 (Estimated)
Dates: Start 2021-09-03 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Choroidal thickness | 30-36 weeks of gestational age
  Choroidal thickness was measured by optical coherence tomography.

SECONDARY OUTCOMES:
Retinal nerve fiber layer thickness | 30-36 weeks of gestational age
  Retinal nerve fiber layer thickness was measured by optical coherence tomography
Retinal vascular density | 30-36 weeks of gestational age
  Percentage of retinal vascular density was measured by optical coherence tomography angiography
Corneal thickness | 30-36 weeks of gestational age
  Corneal thickness was measured by corneal topography

CONTACTS AND LOCATIONS:
Overall Officials: Suthasinee Sinawat, MD, Principal Investigator — KKU Eye Center, Department of Ophthalmology, Faculty of Medicine, Khon Kaen University
Locations (1):
- KKU Eye Center, Faculty of Medicine, Khon Kaen University, Phu Wiang, Changwat Khon Kaen, Thailand